CLINICAL TRIAL: NCT06580639
Title: The Role of a Mycobacterium Growth Inhibition Assay to Quantify Host Immune Control of M. Tuberculosis From Healthy Blood Donors and Patients With Latent or Active Tuberculosis.
Brief Title: The Role of a Mycobacterium Growth Inhibition Assay to Quantify Host Immune Control of M. Tuberculosis
Acronym: MGIA
Status: Recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Thomas Schon, Professor, Linkoeping University
Other Study IDs: 2022-06858-02
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Tuberculosis; Immunologic Activity Alteration
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMCs are collected and frozen in liquid nitrogen. Whole blood is stored separately for DNA and epigenetic analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy Individuals: Patients with a negative IGRA (Quantiferon) who are apparently healthy.
  Interventions: Other: No intervention.
- Close contacts to patients with active TB: Close contacts to patients with active, smear positive pulmonary TB.
  Interventions: Other: No intervention.
- Patients with (latent) tuberculosis infection: Patients without active TB who have a positive IGRA (Quantiferon Plus) result.
  Interventions: Other: No intervention.
- Patients with active TB: Culture or PCR-verified active TB who are initiated on treatment.
  Interventions: Other: No intervention.

INTERVENTIONS:
Other: No intervention. — Blood sampling for analysis of mycobacterial growth inhibition assay (MGIA) analysis.

SUMMARY:
The goal of this observational study is to learn about how the blood leucocytes from patients with and without exposure or disease from tuberculosis (TB) are able to kill live mycobacteria (M. tuberculosis). The main question it aims to answer is:

Is intracellular growth suppression of M. tuberculosis in peripheral blood mononuclear cells variable among healthy blood donors and higher than in patients with latent TB compared to active TB?

DETAILED DESCRIPTION:
Background: The host immune response is crucial in determining the outcome after exposure to Mtb. A substantial proportion of exposed individuals (40-70%) never develop infection indicating an efficient cell mediated immune response against Mtb and early clearance by the host immune defense (Verall et al, Immunology 2014). Thus, the outcome of exposure is highly dependent on host immunity. In this study, our aim was to investigate whether the previously developed mycobacterium groth inhibition assay (MGIA) method (Andersson et al, Tuberculosis 2020) could be used to quantify the host immune response to Mtb.

Study design: In this study we will include healthy donors (n=80), patient with active TB (n=40), subjects recently exposed to active TB (n=80) and patients with latent TB (LTBI) (n=80). Exclusion criteria for all groups are known HIV infection or other immunosuppression from treatment or disease. Patients and healthy blood donors will be recruited at the departments of infectious diseases in Region Kalmar and Region Östergötland. From patients giving oral and written consent, 40 ml of blood will be collected for MGIA analysis.

Primary aim: To determine the difference in MGIA between healthy blood donors and patients with latent and active TB as well as the variation in host control of Mtb within each group.

Method: The Mycobacterial growth inhibition assay (MGIA) using human PBMCs isolated by density gradient by Lymhoprep (Axis-Shield) and SepMate tubes (StemCell Technologies) will be performed as described in study I with minor modifications. The PBMCs are infected with GFP expressing M. tuberculosis H37Rv and intracellular growth of Mtb and viability of PBMCs are assessed by live-cell imaging (Incucyte©) and measured as relative fluorescence units (RFU) during 5 days with and without stimulation with the purified protein derivate (PPD) is included. The cytokine response following exposure to gamma-irradiated H37Rv will be quantified by Olink proteomics.

ELIGIBILITY:
Inclusion Criteria: Healthy blood donors or subjects who will get vaccinated.

Exclusion Criteria:Known HIV infection, not Swedish citizen, chronic liver och kidney disease,immunosuppression from treatment or disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who are attending the infectious disease clinics at region Östergötland och region Kalmar, Sweden.
Sampling Method: Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Mycobacterial inhibition of host macrophages | Up to 10 days incubation
  Mycobacterial inhibition of host macrophages
Mycobacterial inhibition of host peripheral blood mononuclear cells (PBMCs) | Up to 10 days incubation
  Mycobacterial inhibition of host peripheral blood mononuclear cells (PBMCs)

SECONDARY OUTCOMES:
Cytokine expression of host peripheral blood mononuclear cells (PBMCs) | 24 hours
  Proteome analysis following exposure of PBMCs to gamma-irradiated M. tuberculosis

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schoen, Professor, Principal Investigator — Linkoeping University
Locations (2):
- Sweden (2):
  - Kalmar County Hospital, Kalmar
  - Dept of Infectious Diseases, Linköping